CLINICAL TRIAL: NCT06502106
Title: Internet-delivered Trauma-focused Cognitive-behavioral Therapy as an Early Intervention After Sexual Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Traumamottagning Centrum för Sexuell Hälsa, Skånes Universitetssjukhus, Malmö (Unknown)
Responsible Party: Principal Investigator, Maria Bragesjo, Princicpal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01105-01
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Stress Disorder; Post Traumatic Stress Disorder
Keywords: condensed prolonged exposure; PTSD; internetdelivered; trauma; early intervention; prevention; CIPE
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Prolonged exposure will be offered in a brief digital format with therapist support for three weeks. Treatment comprises of psychoeducation, rationales, in vivo exposure, imaginal exposure and relapse prevention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Condensed Internet delivered prolonged exposure (CIPE) (Experimental): Condensed Internet delivered prolonged exposure (CIPE) for three weeks with therapist support.
  Interventions: Behavioral: Condensed Internet delivered prolonged exposure (CIPE)

INTERVENTIONS:
Behavioral: Condensed Internet delivered prolonged exposure (CIPE) — Condensed Internet delivered prolonged exposure (CIPE) with therapist support for three weeks.

SUMMARY:
The research aims to assess the practicality and implementation aspects, effectiveness, and processes of change related to Condensed Internet-delivered Prolonged Exposure (CIPE) administered as an early trauma focused intervention after sexual assault. Eligible participants are individuals seeking help at Traumamottagning Centrum för Sexuell Hälsa, Malmö who have been exposed to sexual assualt in the past two months and exhibit psychological symptoms in response to that.

DETAILED DESCRIPTION:
The study is un-controlled with 30 participants that will undergo a brief trauma-focused Internet-based CBT treatment, delivered as a three-week treatment comprising of four modules (psychoeducation/rational, in vivo exposure, imaginal exposure and relapse prevention). The primary outcome is level of symptoms of post traumatic stress rated by the PCL-5. Secondary outcomes are level of symptoms of post traumatic stress using the Clinician Administered PTSD Scale version 5 (CAPS-5) and The International Trauma Questionnaire (ITQ), level of depression (PHQ-9), quality of life (WSAS and EQ-5D ) dropout rate, rates of inclusion, attrition, adherence,and negative effects.

Qualitative data using a semi-structured interview will be gathered from participants at the end of the treatment collecting data on participants' views on the treatment, preferences for this type of treatment and how to further improve it.

The treatment effects will be evaluated using a within-group design with repeated measurements. Participants in the study will be will recruited from patients treated for sexual assault at Traumamottagning Centrum för Sexuell Hälsa, Malmö.

ELIGIBILITY:
Inclusion Criteria:

* Experienced trauma in the past two months according to criterion A for PTSD in the DSM-5 (exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence).
* At least mild clinical symptoms assessed using the PCL-5 cut-off >10
* ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, borderline personality disorder, high suicidal risk)
* Unable to read and write in Swedish
* Receiving other psychological trauma-focused treatment
* Ongoing trauma-related threat (e.g., living with a violent spouse)
* Not stable dose of antidepressant medication the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, weekly through three weeks of treatment, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Clinician Administered PTSD Scale version 5 (CAPS-5), the gold standard clinical interview to assess PTSD symptom severity and diagnosis of PTSD | Three months after treatment completion.
  The CAPS-5 is a 20-item clinical administered interview based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
The International Trauma Questionnaire (ITQ) | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self- Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in psychosocial impairment measured by The Work and Social Adjustment Scale (WSAS), adapted to symptoms of post-traumatic stress. | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  WSAS is a short, self-reported instrument consisting of five items about psychosocial impairments rated on a nine-point Likert scale. A higher score means more severe impairment.
Change in quality of life measured by EQ-5D | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.
Change in use of alcohol measured by Alcohol Use Disorders Identification Test (AUDIT) | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  point Likert scale (0-4) and differentiates between hazardous alcohol use, dependence symptoms, and harmful alcohol use. The total score of the AUDIT ranges from 0 to 40 points, with a higher score reflecting greater risk of alcohol use disorders.
Change in drug use measured by Drug Use Disorders Identification Test (DUDIT) | Baseline, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  Self-rated questionnaire on drug use. It contains 11 items that are scored on a five-point Likert scale (0-4) and differentiates between hazardous drug use, dependence symptoms, and harmful drug use. The total score of the DUDIT ranges from 0 to 44 points, with a higher score reflecting greater risk of drug use disorders.

OTHER OUTCOMES:
Adverse events related to treatment measured by an openended question | Baseline, weekly through three weeks of treatment, post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  Adverse events related to treatment measured by with a free text option where participant is instructed to describe the possible event in detail. If the participant reported any adverse event, additional follow-up questions about intensity, duration etc. will also be given.
Adverse events realted to treatment measured by Negative effects questionnaire (NEQ) | Post-treatment (immediately after treatment completion at three weeks), and the 1 month, 3 month, 6 month and 12 month follow up.
  Self-rated questionnaire on negative effects. It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.
Participants satisfaction with treatment | Immediately after treatment completion.
  Qualitative questions pertaining participants satisfaction with the treatment.
Participants satisfaction with treatment as measured by the CSQ-8 | Immediately after treatment completion.
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Number of completed treatment modules | Baseline up to 3 weeks
  Data will be gathered on total number of completed modules during the three week treatment.
Number of completed home work assignments by the participant during the treatment period | Baseline up to 3 weeks
  Data will be gathered on total number of completed home work assignments by the participant during the three week treatment.
Number of messages sent and received in the digital platform | Baseline up to 3 weeks
  Data will be gathered on total number of messages sent and received in the digital platform during the three week treatment.
The proportion of participants that conducts the weekly measures and further assessment points | Baseline up to 3 weeks
  The proportion of participants that conducts the weekly measures and further assessment points
The proportion of participants that go through the entire treatment period | Baseline up to 3 weeks
  The proportion of participants that go through the entire treatment period
Number of drop-outs from treatment | Baseline up to three weeks]
  Number of drop-outs from treatment
Rates of inclusion to the study | Baseline
  Data on rates of inclusion will be considered as an indication of the feasibility of the intervention.
Level of perceived socialm support measured by Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, post-treatment (immediately efter treatment completion)and at the 1, 3, 6 and 12-month follow up.
  Self-rated questionnaire on perceived social support. It contains 12 items that are scored on a seven-point Likert scale (1-7) and differentiates between perceived support from family, friends, and a significant other. The total score of the MSPSS ranges from 12 to 84 points, with a higher score reflecting greater perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Traumamottagning Centrum för Sexuell Hälsa, Skånes Universitetssjukhus, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No